CLINICAL TRIAL: NCT00204698
Title: Identification of Molecular Markers of Inflammatory Mediators in Posterior Laryngitis Due to Laryngopharyngeal Reflux and Evolution With PPI Treatment
Brief Title: Laryngopharyngeal Reflux and Proton Pump Inhibitor (PPI) Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Susan Thibeault, Ph.D., University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 11690
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Laryngopharyngeal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): All subjects will be given active drug.
  Interventions: Drug: Aciphex

INTERVENTIONS:
Drug: Aciphex — 20 mg of aciphex taken twice daily

SUMMARY:
This study proposes to investigate prospectively, the presence of molecular markers for inflammation in laryngopharyngeal reflux (LPR) patients and to study the effect of a proton pump inhibitor (Aciphex) on these molecular markers.

The investigators will be evaluating a group of patients before and after treatment. This group will be patients that have untreated laryngopharyngeal reflux diagnosed by laryngoscopic assessment and a 24-hour probe.

DETAILED DESCRIPTION:
Objectives:

This study proposes to investigate prospectively, the presence of molecular markers for inflammation in LPR patients and to study the effect of a proton pump inhibitor on these molecular markers. This study will provide important data regarding the etiology of LPR. It will also provide vital information about the present standard treatment for LPR and why it is not universally successful.

Patient Selection Criteria:

The subject group will consist of 25 subjects who have untreated LPR diagnosed by laryngoscopic assessment and 24-hour pH probe.

Design:

The presence of proinflammatory cytokines will be measured at the gene and protein expression levels from PL biopsies with gene specific semiquantitative reverse transcription-polymerase chain reaction and Western Blot analysis.

Statistical Methods, Data Analysis, and Interpretation:

Null Hypothesis: There will be no difference in cytokine expression in the posterior larynx in patients with laryngopharyngeal reflux after 10 weeks of treatment with Aciphex, a proton pump inhibitor.

Alternative Hypothesis: There will be a difference in cytokine expression in the posterior larynx in patients with laryngopharyngeal reflux after 10 weeks of treatment with Aciphex, a proton pump inhibitor.

Effect size = 30% (based upon review of the literature for cytokines in inflammatory states)

Standard Deviation = 30

Standard Effect Size = effect size/standard deviation = 30/30 = 1

With an alpha of 0.05, power 0.1 (90% power), sample size should be 22. Therefore we have chosen 25 subjects in case of error in molecular studies.

Paired t-tests will be utilized to compare differences between cytokine levels for experimental group initiation and completion of medication.

ELIGIBILITY:
Inclusion Criteria:

* The subject group will consist of 25 subjects who have untreated LPR diagnosed by laryngoscopic assessment and 24-hour pH probe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The presence of proinflammatory cytokines will be measured at the gene and protein expression levels from PL biopsies with gene specific semiquantitative reverse transcription-polymerase chain reaction and western blot analysis. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Thibeault, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Thibeault SL, Smith ME, Peterson K, Ylitalo-Moller R. Gene expression changes of inflammatory mediators in posterior laryngitis due to laryngopharyngeal reflux and evolution with PPI treatment: a preliminary study. Laryngoscope. 2007 Nov;117(11):2050-6. doi: 10.1097/MLG.0b013e318124a992. PMID 17721405